CLINICAL TRIAL: NCT00729313
Title: A Phase III Multicentre Randomised Double-blind Comparative Study of Efficacy and Safety of Lanreotide 30 mg Versus Placebo for Treatment of Patients With Digestive Fistulae
Brief Title: Efficacy and Safety of Lanreotide Versus Placebo for Treatment of Patients With Digestive Fistulae
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Joelle Blumberg, Ipsen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-54-52030-053
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Digestive Fistulae
Keywords: Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug: Lanreotide 30 mg microparticle formulation
  One intra-muscular injection.
  A (maximum) 60 day "treatment" period (6 intra-muscular injections of lanreotide 30 mg microparticle formulation every 10 days): according to the patient's treatment response at 72h
  For non-responders patients lanreotide will be stopped.
  Interventions: Drug: Lanreotide microparticles
- 2 (Placebo Comparator): One intra-muscular injection.
  A (maximum) 60 day "treatment" period (6 intra-muscular injections of placebo every 10 days): according to the patient's treatment response at 72h.
  Non-responder patients having received placebo on the first injection should receive an open-labelled lanreotide treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanreotide microparticles
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of the protocol, is to determine whether lanreotide 30 mg is effective in the treatment of patients with digestive fistulae.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether lanreotide 30mg compared to placebo is effective on the evolution of drainage volume of digestive fistulae in the 72 hours following the beginning of treatment and on the spontaneous closure time of digestive fistulae.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pancreatic, duodenal, or small intestine fistula
* Patient with simple, externalised fistula
* Patient with fistula for which a medical conservative treatment is considered
* Patient with:
* for pancreatic fistulae: a mean drainage volume more than or equal to 100 ml/24h over 48 hours or more than or equal to 50 ml / 24h over 3 days and a concentration of amylase in the drainage fluid 3 times higher than in the serum over at least 2 or 3 consecutive days respectively,
* for duodenal and small intestine fistulae: a mean drainage volume more than or equal to 100ml/24h over 2 days

Exclusion Criteria:

* Patient expected to require a surgical treatment of the fistula during the study
* Patient having uncontrolled intra-abdominal sepsis; Crohn's disease; radiotherapy lesions of the small bowel; a mesenteric vascular insufficiency; a fistula localised in cancer-infiltrated areas; a distal obstruction; an exposed fistula of the small intestine; or intra-abdominal foreign bodies.
* Patient receiving long-term corticotherapy
* Patient having received any somatostatin analogue as curative treatment of the fistula or any PRF somatostatin analogue within the previous month.
* Patient having previously undergone a transplant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2000-04; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with a reduction of fistula drainage volume > 50% of baseline at 72 hours. | Fistula drainage volume on 3rd day.

SECONDARY OUTCOMES:
Closure time of digestive fistulae will be defined by the interval between D0 (day of the first injection) and the date of spontaneous closure of the fistula. | Day 60
Pancreatic or duodenal and small intestine fistula closing rate within D60 | Day 60
Number of injections received by each patient | End of study
Percentage of fistula recurrence during the follow-up period | Duration of follow-up period for each patient is of 1 month
Percentage of mortality in each group | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (19):
- France (17):
  - Hôpital Nord, Amiens
  - CHU J. Minjoz, Besançon
  - Hôpital Avicenne, Bobigny
  - Hôpital de la Cavale Blanche, Brest
  - Hôpital Louis Mourier, Colombes
  - Hôpital Henri Mondor, Créteil
  - Hôpital A. Michallon, Grenoble
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Edouard Herriot, Lyon
  - Hotel Dieu, Lyon
  - Hôpital Nord, Marseille
  - Hôpital Lariboisière, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Pontchaillou, Rennes
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Trousseau, Tours
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- Russia (2):
  - Institute of Surgery n.a. A.V. Vishnevsky, Moscow
  - National Research Centre of Surgery, Moscow

REFERENCES:
- [Result] Gayral F, Campion JP, Regimbeau JM, Blumberg J, Maisonobe P, Topart P, Wind P; Lanreotide Digestive Fistula. Randomized, placebo-controlled, double-blind study of the efficacy of lanreotide 30 mg PR in the treatment of pancreatic and enterocutaneous fistulae. Ann Surg. 2009 Dec;250(6):872-7. doi: 10.1097/sla.0b013e3181b2489f. PMID 19953707